CLINICAL TRIAL: NCT05201846
Title: Effect of Continuous Subcutaneous Insulin Injection in Pediatric Patients With Type 1 Diabetes Using Multiple Daily Insulin Injections
Brief Title: Comparison of CSII and MDI in Pediatric Patients With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Choong Ho Shin, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21111431275
Record Dates: First submitted 2021-12-17; First posted 2022-01-21 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous subcutaneous insulin infusion (Experimental): Continuous subcutaneous insulin infusion using insulin pump (DIA:CONN G8) with continuous glucose monitoring
  Interventions: Device: DIA:CONN G8 insulin pump
- Multiple daily insulin injection (Active Comparator): Multiple daily insulin injection with continuous glucose monitoring
  Interventions: Other: Multiple daily insulin injection

INTERVENTIONS:
Device: DIA:CONN G8 insulin pump — Subjects on continuous subcutaneous insulin infusion system with CGM
  Arms: Continuous subcutaneous insulin infusion
Other: Multiple daily insulin injection — Subjects on multiple daily insulin injection with CGM
  Arms: Multiple daily insulin injection

SUMMARY:
Prospective, randomized, open-label, two-sequence crossover study to investigate the effects of continuous subcutaneous insulin injection (CSII, using DIA:CONN G8 insulin pump) in pediatric patients with type 1 diabetes using multiple daily insulin (MDI) injection

DETAILED DESCRIPTION:
This trial consists of two crossover periods of 5 weeks each (MDI to CSII or CSII to MDI), followed by an extended period of 12 weeks (MDI or CSII). Each intervention period has wash-out period (5 days) excluded from the outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is aged 2-17
2. The subject with one or more of the below at diagnosis

   * serum c-peptide < 0.6 ng/mL
   * positive glutamic acid decarboxylase (GAD) antibody
   * positive Islet cell antibody
   * positive anti-Insulin antibody
   * positive anti-Islet Antigen-2 (IA-2) antibody
3. The subject was diagnosed with type 1 diabetes ≥ 1 year
4. The subject is treated with multiple daily insulin injection
5. The subject must have available continuous glucose monitoring (CGM) data with a percentage of active CGM time ≥ 70% in the past 4 weeks.

Exclusion Criteria:

1. Subjects who were treated with insulin pump therapy within 12 weeks prior to trial
2. Any systemic treatment with drugs known to interfere with glucose metabolism within 12 weeks prior to trial
3. Subjects with underlying hematologic disorders that can affect the HbA1c levels
4. Subjects with underlying medical disorders that can affect glucose metabolism
5. Subjects with a neuropsychiatric disorder such as depression or eating disorder
6. Subjects with underlying thyroid disorders and abnormal thyroid function

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Time in range | 30 days
  glucose level between 70-180 mg/dL derived from continuous glucose monitoring

SECONDARY OUTCOMES:
Time above range | 30 days
  glucose level > 180 mg/dL derived from continuous glucose monitoring
Time below range | 30 days
  glucose level < 70 mg/dL derived from continuous glucose monitoring
Mean sensor glucose | 30 days
  mean sensor glucose level derived from continuous glucose monitoring
Coefficient of variation | 30 days
  Standard deviation * 100 / mean (derived from continuous glucose monitoring)
Glucose management indicator | 30 days
  estimated HbA1c levels derived from continuous glucose monitoring
Glycated albumin | Changes from baseline to after 30 days of intervention
  Glycated albumin level
Quality of life measurements (general) of patients and parents | At the end of intervention (30 days)
  Measured by PedsQL (Pediatric Quality of Life InventoryTM) Generic Core Module 4.0 (values: 0~100, higher score means better outcome)
Quality of life measurements (diabetes-specific) of patients and parents | At the end of intervention (30 days)
  Measured by PedsQL (Pediatric Quality of Life InventoryTM) Diabetes Module 3.0 (values: 0~100, higher score means better outcome)
Children's Depression inventory of patients | At the end of intervention (30 days)
  Measured by Korean Children's Depression Inventory, 2nd Edition (values: 0~100, higher score means worse outcome)
Perceived stress scale of parents | At the end of intervention (30 days)
  Perceived stress scale (values: 0~56, higher score means worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Choong Ho Shin, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul